CLINICAL TRIAL: NCT02800681
Title: Psychopathological Differences Between Asperger Syndrome/Normal IQ, no Language Impairment Autism Spectrum Disorder and Schizotypal Disorder in an Adult Sample
Brief Title: Psychopathological Differences Between Asperger Syndrome and Schizotypal Disorder in an Adult Sample
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: The Danish Autism Centre (Unknown)
Responsible Party: Principal Investigator, Maria Elisabeth Nilsson, MD, PhD-student, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Other Study IDs: E-61120-06
Record Dates: First submitted 2016-05-24; First posted 2016-06-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Asperger Syndrome; Autism Spectrum Disorder; Schizotypal Personality Disorder
Keywords: Asperger Syndrome; Autism Spectrum Disorder; Schizotypal disorder; Schizophrenia Spectrum Disorder; Psychopathology; Examination of Anomalous Self Disorder; Autism Diagnostic Observation Schedule; Phenomenology; Differential diagnosis; Young Adult
MeSH Terms: conditions — Asperger Syndrome; Autism Spectrum Disorder; Schizotypal Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asperger syndrome: 1. Expert panel evaluation for identification of participants with typical symptoms
  2. Semi-structured psychopathological interviews for general psychopathology, psychopathology within the schizophrenia spectrum, and psychopathology within the autism spectrum
  3. Self-administered rating scales for assessment of autistic traits, schizotypal personality and subjective psychological well-being
  4. Other general interviewer ratings for assessing functioning and severity of psychopathology
  Interventions: Other: Expert panel evaluation; Other: Semi-structured psychopathological interviews; Other: Self-administered rating scales; Other: Other general interviewer ratings
- Schizotypal disorder: 1. Expert panel evaluation for identification of participants with typical symptoms
  2. Semi-structured psychopathological interviews for general psychopathology, psychopathology within the schizophrenia spectrum, and psychopathology within the autism spectrum
  3. Self-administered rating scales for assessment of autistic traits, schizotypal personality and subjective psychological well-being
  4. Other general interviewer ratings for assessing functioning and severity of psychopathology
  Interventions: Other: Expert panel evaluation; Other: Semi-structured psychopathological interviews; Other: Self-administered rating scales; Other: Other general interviewer ratings

INTERVENTIONS:
Other: Expert panel evaluation — From the medical records, described social and psychiatric history and observed psychiatric symptoms will be summarized and presented to two senior psychiatric consultants. The panels evaluation ensures the identification of subjects with typical symptoms, according to a best estimate clinical consensus.
  The panel divides the participants into 4 groups: 'participant with symptoms typical of AS', 'participant with symptoms typical of SD', 'participant with inconclusive/non typical symptoms' and 'non eligible participant'.
Other: Semi-structured psychopathological interviews — Included participants are asked for a detailed social and developmental history and interviewed with 3 semi-structured interviews: 1. Schedules for Assessment in Neuropsychiatry (SCAN); Covering psychopathology and behaviour associated with the major psychiatric disorders. 2. Autism Diagnostic Observation Schedule (ADOS), module 4; An assessment to identify symptoms within the autism spectrum. 3. Examination of anomalous self-experience (EASE); A checklist for exploration of experiential anomalies. The Ph.D.-student will obtain social and developmental history and carry out SCAN and EASE interviews. ADOS will be carried out by a consultant psychologist at The Danish Autism Centre.
Other: Self-administered rating scales — 1.The Autism Quotient (AQ), a 50 question scale, for the assessment of autistic traits, 2. The Schizotypal Personality Questionnaire (SPQ), a 74 item scale, for the assessment of schizotypal personality, 3. The WHO-5 Well-Being Index (WHO-5), a 5 item scale, for the assessment of subjective psychological well-being.
Other: Other general interviewer ratings — 1. Global Assessment of Functioning (GAF), a numeric scale (1 through 100) for assessing social, occupational, and psychological functioning, 2. The Clinical Global Impressions scale (CGI-Severity), an assessment of the clinician's global view of the patient's severity of psychopathology on a 7 point scale.

SUMMARY:
The purpose of this study is to identify psychopathology (psychiatric symptoms) that can differentiate between Schizotypal Disorder (SD) and Asperger Syndrome (normal IQ, no language impairment Autism Spectrum Disorder) (AS) in young adults.

With our present knowledge, the differentiation between AS and SD can be difficult, as they both present with social difficulties, odd (but not psychotic) behaviour, and a 'feeling of not being as everyone else'. Studies suggest that adults with AS symptoms are either overlooked, or diagnosed within the schizophrenia spectrum in Adult Psychiatry.

A 'correct' diagnosis is important, as it is the first step towards the most optimal plan, treatment and rehabilitation for the patient. The only way to diagnose psychiatric illness is the description of present psychopathology.

To identify symptoms that can differentiate between the two disorders, we will use semi-structured interviews to explore present psychopathology in young adults with typical symptoms of SD and AS respectively, with special focus on presence of alterations in self-experience. Alterations in self-experience are typical for the schizophrenia spectrum, and are therefore not thought to be equally present in AS and SD.

The hypotheses are that the total level of altered experiences is higher in SD, than in AS, and with a different pattern of altered experiences in SD than in AS. If the hypotheses are true, an examination of altered self-experience will be valuable to aid clinical differentiation between the two disorders.

DETAILED DESCRIPTION:
Background: SD is a non-psychotic disorder within the Schizophrenia Spectrum (in ICD-10), and has a prevalence of 3.9 % in adult samples. Autism Spectrum Disorder (ASD), a pervasive developmental disorder (including AS), has a prevalence of 1 %.

SD is typically diagnosed in young adults, whereas AS typically is diagnosed in childhood. Sometimes however, the AS symptoms first become invalidating in young adulthood, where social demands exceed the individual's capacity. In these cases, patients with symptoms corresponding to AS, might first be diagnosed as young adults. In Adult Psychiatry though, experience with diagnosing ASD is scarce, and studies suggest that adult patients presenting with symptoms corresponding to AS, are either overlooked, or diagnosed within the schizophrenia spectrum.

Psychiatric diagnosis: Description of present psychopathology is the only way to diagnose psychiatric illness. An accurate diagnosis is crucial for a relevant treatment and rehabilitation plan for the individual patient, as the diagnosis guides the help and support offered. Further, to properly guide neuro-psychiatric research, high diagnostic accuracy is imperative. This study will refer to the diagnostic criteria defined in ICD-10, when including participants, as ICD-10 is the principal diagnostic system in Denmark.

Altered self-experience: Alterations in self-experience are considered highly specific for the schizophrenia spectrum, and are therefore not thought to be present in equal amounts and/or distribution in ASD. If this is true, an examination of anomalous self-experiences would be valuable to aid clinical differentiation between SD and AS. For patients with altered self-experience, the experience of him-/herself as a subject is disturbed. This means that the form and structure (rather than content) of the patients' thoughts and experiences is altered.

Aim, objectives and hypotheses: The aim is to do an in depth exploration of differences in present psychopathology (psychiatric symptoms) in young adults with SD and AS. This will elaborate and refine our understanding of SD and AS specifically, and ASD and schizophrenia spectrum disorders in general.

The objectives are to; 1. Explore differences in psychopathology between young adults with SD and AS and, 2. Contribute to both the general and the specific (in SD and AS respectively) description of the autism concept.

The hypotheses are that; 1. The total level of altered experiences (EASE total score) is higher in SD than in AS and, 2. The pattern of most occurring altered experiences (individual EASE items) is different in AS, compared to SD.

Material and methods: The study is observational and comparative in design, and will include 100 participants; 50 diagnosed with SD, and 50 with AS. The included subjects medical history will be revised by two senior psychiatric consultants, ensuring identification of participants with typical symptoms. Further, all included participants will be assessed with three semi-structured psychopathological interviews, general symptom and functional scores and self-reports.

Co-ratings: All study interviews will be videotaped, and a subset of the taped SCAN and EASE interviews will be co-rated within the research group. Co-ratings will also routinely be performed amongst psychologists at The Danish Autism Centre, who conducts the ADOS interviews.

Statistical analyses: To investigate between group differences, group wise comparisons between SCAN algorithms, ADOS algorithms and EASE outcomes will be applied. Further, secondary correlations across psychopathological domains will be explored, and explorative cross-diagnostic factor analysis will be performed.

Ethical considerations: Prior to inclusion a differentiated informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of Asperger syndrome (F84.5) or infantile autism (F84.0) with normal IQ and no language impairments or schizotypal disorder (F21)
* Age 18-30 (both inclusive)

Exclusion Criteria:

* Known non-verbal IQ < 80 (verbal IQ < 70) or an educational level corresponding to <9 years of primary education
* Diagnosed with both Schizophrenia Spectrum Disorder and Autism Spectrum Disorder
* Psychotic symptoms (< 1 day of duration, lifetime)
* Severe physical illness (life-limiting, or limiting interview capacity)
* Organic brain disorder (corresponding to ICD-10 chapter F00-09)
* Active heavy alcohol or substance abuse (corresponding to ICD-10 definitions)
* Not fluent in the Danish language
* Forensic patients

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Only already diagnosed participants are recruited, from specialised units. This is essential, as inclusion of participants with typical symptoms, reduces confounding of the results by diagnostic uncertainty.
  Participants with SD will be recruited from OPUS-teams (a specialized treatment program for patients with first episode of schizophrenia spectrum disorder), within the Mental Health Services in the Capitol Region of Denmark, and participants with AS from The Danish Autism Centre (a non-profit organization for people with ASD).
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Level of altered experiences | Assessed within 1,5 years from study inclusion start
  Total score, Examination of Anomalous Self Experience (EASE)
Pattern of most occurring altered experiences | Assessed within 1,5 years from study inclusion start
  Pattern of individual items, Examination of Anomalous Self Experience (EASE)

SECONDARY OUTCOMES:
Autism Spectrum symptom load | Assessed within 1,5 years from study inclusion start
  Total score, Autism Diagnostic Observation Schedule (ADOS), module 4
Schizophrenia Spectrum symptom load | Assessed within 1,5 years from study inclusion start
  Score, Schedules for Assessment in Neuropsychiatry (SCAN)
Self-reported Autism Spectrum symptom load | Assessed within 1,5 years from study inclusion start
  Score, The Autism Quotient (AQ)
Self-reported Schizotypia symptom load | Assessed within 1,5 years from study inclusion start
  Score, Schizotypal Personality Questionnaire (SPQ)
Self-reported well-being | Assessed within 1,5 years from study inclusion start
  Score, World Health Organization Well-Being Index (WHO-5)

OTHER OUTCOMES:
Global severity of symptoms assessment | Assessed within 1,5 years from study inclusion start
  Score, Clinician Global Impressions Scale (CGI)
Global functioning assessment | Assessed within 1,5 years from study inclusion start
  Score, Global Assessment of Functioning (GAF)

CONTACTS AND LOCATIONS:
Overall Officials: Sidse Arnfred, MD, dr.med., Study Chair — Mental Health Services, Region Zealand, Denmark; Peter Handest, MD, Ph.d., Study Chair — Mental Health Services, the Capitol Region, Denmark
Locations (2):
- Denmark (2):
  - Mental Health Centre Ballerup, Mental Health Services, The Capitol Region, Copenhagen, Ballerup Municipality, Copenhagen
  - The Danish Autism Centre, Herlev

IPD SHARING:
Plan to Share IPD: No